CLINICAL TRIAL: NCT03223389
Title: Effects of Fat Metabolites on Gut Hormone Secretion After Gastric Bypass Surgery
Brief Title: Fat Metabolites and Gut Hormones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Christoffer Martinussen, Medical doctor, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CM-FAT-17
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Overweight and Obesity; Type 2 Diabetes; Bariatric Surgery; Gut Hormones; Dietary Fat
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — tricaprylin; Olive Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 gastric bypass operated patients (Experimental): 3 different oils ingested at separate study days will be tested against each others ability to induce gut hormone secretion.
  Interventions: Dietary Supplement: C-8 dietary oil; Dietary Supplement: Tricaprylin; Dietary Supplement: Olive oil
- 10 healthy control subjects (Experimental): 3 different oils ingested at separate study days will be tested against each others ability to induce gut hormone secretion.
  Interventions: Dietary Supplement: C-8 dietary oil; Dietary Supplement: Tricaprylin; Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: C-8 dietary oil — Ingestion of 13.15 g C-8 dietary oil providing 0.0216 mol of triglycerides.
Dietary Supplement: Tricaprylin — Ingestion of 10.17 g tricaprylin providing 0.0216 mol of triglycerides.
Dietary Supplement: Olive oil — Ingestion of 19 g olive oil providing 0.0216 mol of triglycerides.

SUMMARY:
To investigate the effects of different fat metabolites on gut hormone secretion in gastric bypass operated subjects and BMI-matched controls.

DETAILED DESCRIPTION:
Dietary triglycerides are hydrolyzed during digestion to two fatty acids and one 2-monoacyl glycerol. The study will investigate the effects of these different fat components on gut hormone secretion in gastric bypass operated patients and non-operated BMI-matched controls.

ELIGIBILITY:
Gastric bypass operated patients:

Inclusion Criteria:

* Uncomplicated gastric bypass surgery performed minimum 12 months prior to study

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus prior to or after gastric bypass surgery
* Pregnancy or breastfeeding
* Haemoglobin levels below 6,5 mM
* Gall bladder removal

Healthy control subjects:

Exclusion Criteria:

* Bariatric surgery or complicated upper abdominal surgery
* Gall bladder removal
* Pregnancy or breastfeeding
* Haemoglobin levels below 6,5 mM
* Co-morbidities or medicine significantly affecting glucose metabolism or appetite regulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Within group difference in glucagon-like peptide-1 (GLP-1) secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Comparison of the GLP-1 responses (evaluated by AUC above basal) induced by the different oils.
Within group difference in Gastric Inhibitory Peptide (GIP) secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Comparison of the GIP responses (evaluated by AUC above basal) induced by the different oils.
Within group difference in cholecystokinin (CCK) secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Comparison of the CCK responses (evaluated by AUC above basal) induced by the different oils.

SECONDARY OUTCOMES:
Between group comparison of GLP-1 secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  GLP-1 secretion (evaluated by AUC above basal) in gastric bypass operated patients compared to BMI-matched control subjects for each of the oils.
Between group comparison of GIP secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  GIP secretion (evaluated by AUC above basal) in gastric bypass operated patients compared to BMI-matched control subjects for each of the oils.
Between group comparison of CCK secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  GIP secretion (evaluated by AUC above basal) in gastric bypass operated patients compared to BMI-matched control subjects for each of the oils.
Responses (evaluated by AUC above basal) of insulin within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of C-peptide within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of peptide YY (PYY) within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of oxyntomodulin within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of glucagon within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of bile acids within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of fibroblast growth factor 19 (FGF-19) within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of lipid metabolites (triglyceride, cholesterol, fatty acids) within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of neurotensin within and between groups. | 0-240 min following fat ingestion.
Responses (evaluated by AUC above basal) of glucose within and between groups. | 0-240 min following fat ingestion.
Between group comparison of differences in GLP-1 secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Differences in GLP-1 secretion (evaluated by AUC above basal) induced by the different oils in gastric bypass operated patients compared with differences in BMI-matched control subjects.
Between group comparison of differences in GIP secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Differences in GIP secretion (evaluated by AUC above basal) induced by the different oils in gastric bypass operated patients compared with differences in BMI-matched control subjects.
Between group comparison of differences in CCK secretion (evaluated by AUC above basal). | 0-240 min following fat ingestion.
  Differences in CCK secretion (evaluated by AUC above basal) induced by the different oils in gastric bypass operated patients compared with differences in BMI-matched control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Endocrinology, Hvidovre, Denmark

REFERENCES:
- [Derived] Martinussen C, Dirksen C, Bojsen-Moller KN, Svane MS, Carlsson ER, Hartmann B, Clausen TR, Veedfald S, Kristiansen VB, Rehfeld JF, Hansen HS, Holst JJ, Madsbad S. Intestinal sensing and handling of dietary lipids in gastric bypass-operated patients and matched controls. Am J Clin Nutr. 2020 Jan 1;111(1):28-41. doi: 10.1093/ajcn/nqz272. PMID 31742316